CLINICAL TRIAL: NCT04378985
Title: Developing Health Care Service System Based on Participatory Big Data
Brief Title: Developing Health Care Service System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Ji-Won Lee, Professor,Yonsei University College of Medicine,, Gangnam Severance Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 3-2019-0226
Record Dates: First submitted 2020-04-29; First posted 2020-05-07 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wearing a wearable device (the smart watch) for 8 weeks (Experimental): The smart watch to be used in this study is Fitbit Inspire HR. This is a device that has a high worldwide use rate and has active research on its accuracy. It is worn like a normal watch, and it can check heart rate, exercise level, energy consumed, and sleep quality. The values can be checked in real-time on a smartphone application.
  Interventions: Device: Wearing a Wearable device (Fitbit inspire HR)

INTERVENTIONS:
Device: Wearing a Wearable device (Fitbit inspire HR) — 'Wearing a wearable device (the smart watch) for 8 weeks
  The smart watch to be used in this study is Fitbit Inspire HR. This is a device that has a high worldwide use rate and has active research on its accuracy. It is worn like a normal watch, and it can check heart rate, exercise level, energy consumed, and sleep quality. The values can be checked in real-time on a smartphone application.'

SUMMARY:
"Increased health risks and diseases are believed to be caused by multilevel interactions of genetic and environmental factors (including lifestyle habits). Considering the recent advancements in genetic analysis, wearable devices, and big data analysis techniques, collecting and analyzing personal genetic information, lifelogs, and environmental data and predicting the exact health risks of individuals could be possible.

DETAILED DESCRIPTION:
These changes enable the development of healthcare solutions that allow users to actively engage in healthcare and provide appropriate care measures to sufficiently delay or prevent chronic diseases, thereby minimizing the financial losses of the individuals and the society. In particular, chronic diseases such as metabolic syndrome can be prevented or delayed through healthy lifestyle habits. Controversy regarding the effectiveness of using wearable devices and mobile health applications for maintaining lifestyle habits and losing weight exists. Additionally, a study assessing the health of the participants and the disease prevention care for the participants using the genetic data and the lifelog data by the wearable device has not been conducted yet. Therefore, the objective is to operate a lifestyle correction program for examinees who visited a family medicine and health checkup center to develop a user-participation health and disease prevention care system using genetic data and lifelog data. From adults who visited a family medicine and health checkup center, the following should be performed: (1) collect a variety of clinical information, including lifestyle data, physical information, metabolic parameters, genetic information, and metagenomes, which can affect chronic diseases; (2) establish a service model that combines lifestyle data, examination data, and genetic data and analyzes and identifies one's health level through a smartphone application; and (3) examine the effects on the metabolic parameters, lifestyle data, and metagenome (gut microbiome) after using the device (smart healthcare).This pilot study aimed to provide personalized "my data" by linking clinical data and personal lifestyle patterns of the participants who visited a family medicine and examination center.

From adults who visited a family medicine and health check-up center, the following should be performed:

1. Collect a variety of clinical information, including lifestyle data, physical information, metabolic parameters, genetic information, and metagenomes, which can affect chronic diseases
2. Establish a service model that combines lifestyle data, examination data, and genetic data and analyzes and identifies one's health level through a smartphone application
3. Examine the effects on the metabolic parameters, lifestyle data, and metagenome (gut microbiome) after using the device (smart healthcare) "

ELIGIBILITY:
Inclusion Criteria:

1. Korean adults aged between 20 and 65 years who visited a family medicine and health checkup center
2. Individuals who understand and are fluent in Korean language
3. Individuals who provided consent for inclusion in the study
4. Individuals who can complete the study without participating in other intervention studies (medicine, diet, exercise) during the whole research duration
5. Individuals who have no restrictions on their participation in physical activities during the whole research duration

Exclusion Criteria:

1. Individuals who did not provide consent for inclusion in the study or individuals who did not provide complete data
2. Individuals with cognitive dysfunction or inability in using wearable devices
3. Individuals with history of infectious brain diseases, head trauma, thyroid diseases, and substance abuse
4. Individuals with vision, hearing, and speech impairments that can affect examinations
5. Individuals considered unfit to participate in this study by researchers
6. Individuals who do not use smartphones

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Estimated)
Dates: Start 2019-12-20 (Actual); Primary Completion 2021-10-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in metabolic parameter (HOMA-IR) at 8 weeks after smart healthcare intervention | 8 weeks after smart healthcare intervention
  Changes in HOMA-IR (calculated using fasting glucose and insulin level) at 8 weeks after smart healthcare intervention.

SECONDARY OUTCOMES:
Changes in other metabolic parameters, inflammatory parameters, metagenome related to the gut microbiome, and sleep quality, diet, and exercise at 8 weeks after smart healthcare intervention | 8 weeks after smart healthcare intervention
  Changes in lipid profile (total cholesterol, TG, LDL-C, HDL-C levels) at 8 weeks after smart healthcare intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Gangnam Severance Hospital, Seoul, South Korea